CLINICAL TRIAL: NCT00000438
Title: Naltrexone Treatment for Alcoholism: Predicting Outcome
Brief Title: Naltrexone Treatment for Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Mary E. McCaul, Ph.D., Professor, Johns Hopkins University
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIAAAMCC11855; R01AA011855 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: naltrexone (Revia)

SUMMARY:
This study will evaluate the effectiveness of the medication naltrexone (Revia) for treating alcoholism. Individuals will be inpatients for a 2 week period and provide assessments of their alcohol withdrawal symptoms, craving, and mood. Following hospital discharge, individuals will be assigned randomly to receive naltrexone daily, naltrexone twice a day or a placebo. This part of the study will last 12 weeks, with regular measurements of drinking level, craving and mood. Assessments will be conducted 6 and 12 months after the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence.
* Committed to alcohol abstinence as a treatment goal.
* Individuals will be required to identify two family members or close friends who are knowledgeable about their location, drinking behavior, and psychosocial status.

Exclusion Criteria:

* Meets criteria for any other psychoactive substance use disorder (excluding nicotine and caffeine).
* Meets criteria for a major psychiatric disorder and are in need of or currently undergoing pharmacotherapy.
* Females who are pregnant, lactating, or not using a reliable method of contraception.
* Currently experiencing a serious medical condition that would place them at risk or interfere with study participation.
* Experiencing acute hepatitis or liver failure or whose liver function test is more than 3 times normal.
* Have a history of severe allergies, multiple adverse drug reactions or known allergy to naltrexone.
* Vocabulary below the 5th grade reading level.
* Abnormal MRI scan.
* HIV infection due to the neurological sequelae.
* Significant central nervous system diseases.
* Seizure disorder or history of closed head trauma.
* Neuroendocrine disorders.
* Treatment with opiates within the last six months.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192
Dates: Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States